CLINICAL TRIAL: NCT03622983
Title: Cohort of Patients With Pelvic Gynecological Cancer: Constitution of a Collection of Biological Samples With Radioclinical Characterization
Acronym: PELVIMASS2
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: PELVIMASS2; 2016-A00613-48 (Other: ID-RCB)
Record Dates: First submitted 2018-08-01; First posted 2018-08-09 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Pelvic Neoplasms; Endometriosis
MeSH Terms: conditions — Pelvic Neoplasms; Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biomarkers and tumoral samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Collection of sample and data: Collection of biological samples and clinical data
  Interventions: Other: collection of sample and data

INTERVENTIONS:
Other: collection of sample and data — Recovery of surgical waste during surgery planned in the current care and clinical data collection

SUMMARY:
The management of pelvic gynecological cancers (PGC) is based on the determination of extension to guide treatments. The biology of the CGP is constantly evolving and personalized medicine adapted to this biology is currently in full development. For example, sequencing ovarian tumors can select patients who can benefit from anti-PARP therapy. There is therefore a need for patients to have biological samples of their tumor. Various studies on ovarian, endometrial and cervical cancer have sought to identify the factors predictive of recurrence of these cancers. The results obtained are very promising. This study will permit to collect biological samples and detailed clinical data that would allow to test hypotheses and develop a personalized medicine based on clinical and biological characteristics of patients.

DETAILED DESCRIPTION:
The management of pelvic gynecological cancers (PGC) is based on the determination of the extension in order to guide the treatments. The biology of PGC is constantly evolving and personalized medicine adapted to this biology is currently in full development. For example, sequencing of ovarian tumors allows selection of patients who may benefit from anti-PARP therapy. There is therefore a need for patients to have biological samples of their tumor. Various studies on ovarian, endometrial and cervical cancer have sought to identify factors that predict recurrence of these cancers. The results have obtained are very promising, but if coordinator team have at our disposal fundamental and translational data related to the prognosis of PGCs, the coordinator team lack access to a biological collection of these cancers that would allow us to test our hypotheses and to develop personalized medicine related to the clinico-biological characteristics of the patients.

Endometriosis is the 1st cause of chronic pelvic pain (25-40% of women suffering during sexual intercourse) and represents the 1st cause of school and work absenteeism. Unfortunately, it is under-diagnosed and too often inappropriately managed. It is considered that 10 to 15% of the female population of reproductive age has endometriosis. This incidence reaches 50% in women with infertility. There are many similarities between deep endometriosis and pelvic cancers, whether on a physiopathological, epidemiological or clinical level. There are therefore many similarities in the surgical management as well as in the research strategies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pelvic gynecological cancer posed on initial histological analysis or during recurrence;
* Or diagnosis of endometriosis on histology or imaging
* Age ≥ 18 years;
* Affiliation to the general social security scheme;
* Consent signed.

Exclusion Criteria:

* Refusal of the patient;
* Non-affiliation to the general social security scheme.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pelvic gynecological cancer or with endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2037-08 (Estimated)

PRIMARY OUTCOMES:
circulating tumor and DNA | 2 years
Endometriosis tumor and DNA | 2 years

SECONDARY OUTCOMES:
circulating tumor DNA | 5 years
circulating tumor DNA | 10 years
circulating Micro RNA | 2 years
circulating Micro RNA | 5 years
circulating Micro RNA | 10 years
circulating cytokines | 2 years
circulating cytokines | 5 years
circulating cytokines | 10 years
Tumoral DNA | day of surgery

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHI Creteil, Créteil
  - CHU Tenon, Paris

IPD SHARING:
Plan to Share IPD: No